CLINICAL TRIAL: NCT05808062
Title: The Effect of Different Canal Dryness Protocols on the Quality of Matched Single Cone Obturation: A Randomized Clinical Trial
Brief Title: The Effect of Canal Dryness on the Quality of Obturation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, shehabeldin saber, Pofessor, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-038
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Obturation
MeSH Terms: conditions — Bites and Stings | interventions — Root Canal Obturation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total dryness (Active Comparator): matching paper points are used till they come out completely dry
  Interventions: Procedure: Root canal obturation
- Partial dryness (Active Comparator): a single matching cone is inserted in the canal for 3 seconds only.
  Interventions: Procedure: Root canal obturation

INTERVENTIONS:
Procedure: Root canal obturation — Root canal dryness

SUMMARY:
The goal of this clinical trial is to evaluate root canal obturation quality. The questions to answer are

* what is the best protocol for canal dryness before obturation ?
* Is compaction necessary ? Volunteer participants will perform root canal treatment in teeth planned for extraction due to orthodontic reasons

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females (Category: American Society of Anesthesiologists class 1)
* aged 23-25 years
* presenting with sound maxillary premolars (non-carious and not previously restored)
* a radiographically visible root canal outline

Exclusion Criteria:

* dental students of any level were not eligible to avoid including vulnerability factors.
* pregnant volunteers
* volunteers with complicating systemic disease (ASA 3-6)
* poor oral hygiene
* periodontal disease (probing depth >3 mm) related to the tooth

Ages: 23 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
obturation quality | after 30 days
  percentage of voids within the filling by micro CT analysis

CONTACTS AND LOCATIONS:
Overall Officials: Shehabeldin Saber, phD, Principal Investigator — Faculty of Dentistry, The British University in Egypt
Locations (1):
- Faculty of Dentistry, The British University in Egypt, Cairo, El-Sherouk, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after study completion
Access Criteria: PI email

REFERENCES:
- [Result] Zavattini A, Knight A, Foschi F, Mannocci F. Outcome of Root Canal Treatments Using a New Calcium Silicate Root Canal Sealer: A Non-Randomized Clinical Trial. J Clin Med. 2020 Mar 13;9(3):782. doi: 10.3390/jcm9030782. PMID 32183124
- [Derived] Nawar NN, Elashiry MM, El Banna A, Saber SM, Schafer E. Ex-vivo evaluation of clinically-set hydraulic sealers used with different canal dryness protocols and obturation techniques: a randomized clinical trial. Clin Oral Investig. 2024 Oct 27;28(11):612. doi: 10.1007/s00784-024-06006-5. PMID 39463194